CLINICAL TRIAL: NCT00363623
Title: Comparison of Contact Lens Maintenance Systems for Silicone Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: CIBA VISION (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H06 009
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2007-02

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

INTERVENTIONS:
Device: Silicone hydrogel contact lens

SUMMARY:
The primary purpose of this study is to investigate the performance of contact lens maintenance systems when used with silicone hydrogel contact lenses during daily wear over a period of 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Is correctable to at least 20/40 distance visual acuity in each eye with spherical contact lenses.
* Is an experienced soft contact lens wearer for at least 1 month.
* Has no clinically significant anterior eye findings.
* Has no other active ocular disease.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Eye surgery or injury within 12 weeks prior to enrolment.
* Has any systemic disease or ocular abnormality that might interfere with contact lens wear
* Has any pre-existing ocular irritation that would preclude contact lens fitting.
* PMMA lens wear previous 6 months.
* EW or CW in previous 1 month.
* Hydrogen peroxide users
* Latex sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2006-08; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lakkis, BScOptom, PhD, Principal Investigator — Clinical Vision Research Australia, University of Melbourne
Locations (1):
- Clinical Vision Research Australia, Carlton, Victoria, Australia